CLINICAL TRIAL: NCT04571411
Title: Severity of Scorpion Sting in Relation to Hematological Parameters
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sarah Osama Mohamed, Resident Doctor, Assiut University
Other Study IDs: scorpion sting in children
Record Dates: First submitted 2020-09-25; First posted 2020-10-01 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Scorpion Stings
MeSH Terms: conditions — Scorpion Stings

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: CBC — The aim of this study is to investigate the relationship between severity of envenomation and hematological parameter by detectig initial mean platelet volume (MPV), neutrophil/lymphocyte ratio (NLR) and platelet/lymphocyte ratio (PLR) in pediatric patients presenting with a scorpion sting.

SUMMARY:
The aim of this study is to investigate the relationship between severity of envenomation and hematological parameter by detectig initial mean platelet volume (MPV), neutrophil/lymphocyte ratio (NLR) and platelet/lymphocyte ratio (PLR) in pediatric patients presenting with a scorpion sting.

DETAILED DESCRIPTION:
Scorpion stings are common emergency events in many parts of the world. It is common in tropical and subtropical regions. In our locality, Upper Egypt, scorpions still represent and a life hazard, especially to children .The clinical manifestations of scorpionism are due to complex interactions between sympathetic and parasympathetic stimulation.This leads to increased release of neurotransmitters and mediators, resulting in a cascade of pathological events, involving the nervous system, the cardiovascular and the respiratory system, eventually leading to death.Scorpionism results in hormonal and biochemical changes with significant release of catecholamines, increased angiotensin II and inhibition of insulin secretion .The symptoms and signs of envenomation are usually more severe in children, especially younger ones. Local pain represent 66 to 90 percent of stings which is practically immediate, of varying intensity ranging from mild to very intense. It is characterized by tingling, burning, or stinging. Regardless of the severity of envenoming, pain and paresthesia may persist at the site or at the affected limb for several days .Systemic effects become apparent in 10 to 33 percent of patients.After envenomation, symptoms may begin immediately and typically progress to maximum severity within 5 hours. The clinical effects of stings are characterized, cardiovascular, neurological and gastrointestinal effects .Cardiovascular effects are atrial tachycardia, ventricular extrasystoles, T-wave inversion, ST-T wave changes, bundle-branch block. Catecholamine-induced myocarditis and myocardial ischemia results in pulmonary edema and cardiogenic shock.Cardiovascular effects are atrial tachycardia, ventricular extrasystoles, T-wave inversion, ST-T wave changes, bundle-branch block. Catecholamine-induced myocarditis and myocardial ischemia results in pulmonary edema and cardiogenic shock..Gastrointestinal effects: are vomiting, abdominal pain and diarrhea. Also acute pancreatitis has been reported.Cardiovascular toxic effects and acute pulmonary edema are the most important complications of scorpion stings and the most frequent cause of death in the first 24 hours after the sting .Gastrointestinal effects: are vomiting, abdominal pain and diarrhea. Also acute pancreatitis has been reported.Cardiovascular toxic effects and acute pulmonary edema are the most important complications of scorpion stings and the most frequent cause of death in the first 24 hours after the sting .

ELIGIBILITY:
Inclusion Criteria:

* a) Patients presented with scorpion sting

Exclusion Criteria:

* All other envenomation or intoxications

Ages: 0 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: study on children stung by scorpion
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
The aim of this study is to investigate the relationship between severity of envenomation and hematological parameter | baseline
  All patient will be conducted to:
  1. full history including: (Age, gender, weight, time and date of presentation
  2. Full examination including : local
  General Cardiac examination Chest examination

CONTACTS AND LOCATIONS:
Overall Officials: Yasser Gamal Abl Elrahman, lecture, Principal Investigator — Assiut University

REFERENCES:
- [Result] Adiguzel S, Ozkan O, Inceoglu B. Epidemiological and clinical characteristics of scorpionism in children in Sanliurfa, Turkey. Toxicon. 2007 May;49(6):875-80. doi: 10.1016/j.toxicon.2006.12.012. Epub 2007 Jan 10. PMID 17286998
- [Result] Shamoon Z, Peterfy RJ, Hammoud S, Khazaeni B. Scorpion Toxicity. 2023 Aug 8. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK430928/ PMID 28613678
- [Result] Chippaux JP. Estimating the global burden of snakebite can help to improve management. PLoS Med. 2008 Nov 4;5(11):e221. doi: 10.1371/journal.pmed.0050221. PMID 18986211
- [Result] Ahmed AE, Abdel-Baseer KA, Saad K, Hassan AF, El-Houfey AA. Endocrinological and biochemical changes of scorpionism in children in Upper Egypt. Ther Adv Endocrinol Metab. 2015 Oct;6(5):210-6. doi: 10.1177/2042018815593034. PMID 26445643
- [Result] Ait Laaradia M, El Hidan MA, Marhoume F, Bouimeja B, Oufquir S, Sokar Z, Boumezzough A, Chait A. Buthus lienhardi venom and pathophysiological effects at the histological, hematological, biochemical and motor skills levels. Toxicon. 2018 May;146:106-113. doi: 10.1016/j.toxicon.2018.03.001. Epub 2018 Mar 9. PMID 29526539
- [Result] Horoz OO, Yildizdas D, Aslan N, Gokay SS, Ekinci F, Erdem S, Haytoglu Z, Sertdemir Y, Yilmaz HL. Is there any relationship between initial hematological parameters and severity of scorpion envenomation? Turk J Pediatr. 2020;62(3):394-404. doi: 10.24953/turkjped.2020.03.006. PMID 32558413
- [Result] Cupo P. Clinical update on scorpion envenoming. Rev Soc Bras Med Trop. 2015 Nov-Dec;48(6):642-9. doi: 10.1590/0037-8682-0237-2015. PMID 26676487
- [Result] Chippaux JP. Management of scorpion stings in Africa and the Mediterranean region. Med Sante Trop. 2016 May 1;26(2):130-3. doi: 10.1684/mst.2016.0571. PMID 27412972